CLINICAL TRIAL: NCT07223450
Title: Physiologically Based Pharmacokinetic Modelling of Oral and Intranasal Formulations of Oxycodone in Healthy Volunteers
Brief Title: A Study on Oral and Intranasal Forms of Oxycodone in Healthy Volunteers Using Pharmacokinetic Modeling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-515461-34-00; 2024-515461-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-09; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-06

CONDITIONS: Physiologically Based Pharmacokinetic; Healthy Volunteers
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral oxycodone (Active Comparator)
  Interventions: Drug: oxycodone
- intranasal oxycodone (Experimental)
  Interventions: Drug: Oxycodone IN

INTERVENTIONS:
Drug: Oxycodone IN — 0.1 mg/kg intravenously oxycodone solution administered intranasally
  Arms: intranasal oxycodone
Drug: oxycodone — oral solution 0.1 mg/kg
  Arms: Oral oxycodone

SUMMARY:
This is a single-dose, 2-period, 2-sequence, fasting, open label, crossover randomized design, comparing the pharmacokinetics (PK) and pharmacodynamics (PD) of intranasal and oral oxycodone solutions. The aim will be to characterize the PK and PD of two formulations of oxycodone (intranasal and oral) in healthy subjects, which will be used to verify/validate nasal-CNS-PBPK (Physiologically Based Pharmacokinetic) model predictions following intranasal dosing. A total of 8 healthy male/female subjects will be randomly assigned to one of two sequences in the crossover study. All subjects will receive the same dosage of oxycodone intranasal or oral and the sequence will be determined following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers according to physical examination, vital signs (blood pressure, heart rate and body temperature), ECG and safety laboratory parameters and results should be within normal ranges or considered as non-clinically relevant by the investigator.
* Age ≥ 18 and ≤ 55 years.
* Body weight up to 90 kg
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Able/willing to be compliant with the study restrictions
* Able to read Spanish and adhere to study requirements.
* Signed informed consent prior to any study-mandated procedure.
* Prior therapeutic or recreational experience with opioids (i.e., tramadol, oxycodone, or buprenorphine)

Exclusion Criteria:

* Life-time (current and/or history of) substance use disorders (SUD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Use of any illegal drug within 30 days of screening and throughout participation in the study
* History of smoking or use of nicotine containing products within 3 months of screening and throughout participation in the study
* No acute, chronic, or allergic rhinitis
* Ongoing gastrointestinal diseases or history of gastrointestinal surgery affecting absorption.
* History of severe bronchial asthma or chronic obstructive pulmonary disease,
* Any anatomical abnormality or pathological condition of the nasal cavity based on medical history.
* History of hypothyroidism.
* Subjects with a clinically relevant disease or condition that in the judgment of the investigator might interfere with the safety or subject's ability to comply with study procedures or requirements and/or bias the interpretation of the study results and/or jeopardize the subject's safety.
* Current mental diseases that require prescription drugs.
* Any ophthalmologic condition that could interfere with pupillometry
* Being under any administrative or legal supervision.
* Pregnancy and breastfeeding
* Positive blood or urine test for drugs of abuse or alcohol breath test prior to study drug administration.
* Current and/or history of anxiety or depression not completely recovered within 12 months prior to study drug administration, as assessed by the Dual Diagnosis Screening Interview (DDSI).
* CYP2D6 poor or ultrarapid metabolizers.
* Any clinically relevant findings in physical examination, vital signs, 12-lead ECG and safety laboratory parameters.
* Positive hepatitis or HIV tests (Ag VHB, IgG VHC, Ac VIH).
* Known hypersensitivity to any drug or drug excipients.
* Use of drugs known to induce or inhibit hepatic drug metabolism (check drugs in Appendix 6) within one month prior to study administration or during the study and use of citrus juice during the study.
* Use of sedative medicines such as benzodiazepines or related drugs in the last 3 months.
* Any prescription or over-the-counter (OTC) product, not including oral contraceptives but including analgesics (paracetamol), aspirin, herbal, homeopathic, vitamins, minerals and nutritional supplements within one week prior to study drug administration.
* Intake of foods or beverages containing xanthine (more than 5 cups of coffee, tea or 5 bottles/cans cola drinks) per day.
* Donation of blood or plasma within two months prior to study drug administration
* Transfusion of blood or plasma for medical/surgical reasons in the past 120 days.
* Current or history of inadequate venous access and/or experience of difficulty donating blood.
* Subject included in a clinical trial within 3 months prior to study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
AUC(0-24h) | up to 24 hours
  Area under the curve from 0 time to the last measurable concentration (of intranasal and oral oxycodone), calculated from individual plasma PK concentrations.
Tmax | Blood samples were taken pre-dose and up to 24 hours after start of each Dose
  Time of maximum observed concentration (of intranasal and oral oxycodone), calculated from individual plasma PK concentrations.
Cmax | Blood samples were taken pre-dose and up to 24 hours after start of each Dose
  The mean maximum observed concentration (of intranasal and oral oxycodone), calculated from individual plasma PK concentrations

SECONDARY OUTCOMES:
Treatment-emergent adverse events | from Day 1 to end of study (EOS)
  Treatment-emergent AEs, including potentially clinically significant abnormalities.

OTHER OUTCOMES:
Pupil size | up to 24 hours
  To assess the effects of oxycodone on Pupil size

CONTACTS AND LOCATIONS:
Overall Officials: Rafael De la Torre, PhD, Principal Investigator — Hospital del Mar Research Institute Barcelona
Locations (1):
- Hospital del Mar Research Institute, Barcelona, Spain